CLINICAL TRIAL: NCT04320524
Title: Mixed Methods (Quantitative, Qualitative) Feasability Study Assessing Engagement With the TARA Working Prototype [Version 2] (a Digital Behaviour Change Intervention, DBCI) and Effects of TARA on Behavioural Targets and Medication Adherence in Individuals With COPD
Brief Title: TARA Working Prototype [Version 2]: Feasibility Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Covid, the study could not be initiated as planned.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 0352-2134
Record Dates: First submitted 2020-03-15; First posted 2020-03-25 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental)
  Interventions: Device: Technology-Assisted Respimat Adherence Digital Behaviour Change Intervention

INTERVENTIONS:
Device: Technology-Assisted Respimat Adherence Digital Behaviour Change Intervention — 3 weeks

SUMMARY:
TARA is a Digital Behaviour Change Intervention (DBCI) for Individuals with COPD (IwCOPD), which has been designed using a Human-Centred Design (HCD) methodology. HCD involves, among other elements, members of the target audience in evaluations at multiple stages within the design process.

This feasibility study is primarily designed to assess the acceptability of the DBCI test asset to the target audience. Acceptability as defined for the purpose of this study includes usability of the system, and perceived value and desirability to the end-user audience. As such, engagement in this context is deemed to mean the degree to which the test asset provides a usable, acceptable, desirable and valuable experience to its users during a time-limited trial.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written electronic informed consent (e-consent) in accordance with ICH-GCP and local legislation prior to admission to the study
* Male or female patients
* All patients must have a self-reported confirmation of a physician diagnosis of COPD (or chronic bronchitis or emphysema)
* Age ≥ 40 years
* Patients must be current or ex-smokers
* Modified Medical Research Council (mMRC) Score ≥ 2 (i.e. evidence of activity-related breathlessness)
* Patients must have a current prescription for either Spiriva Respimat or Stiolto Respimat in keeping with their approved labels as well as a short-acting bronchodilator ("rescue medication") for at least 3 months prior to study enrolment
* Participants must be willing to use a smart watch and be willing to complete all data collection requirements (within TARA plus phone interview plus on-line questionnaires)
* Patients must confirm that their treating physician has been informed about their participation in the study (prior to TARA log-in)
* Fluency in written English
* Currently residing in US (for duration of study)
* Participants should be not fully adherent to once daily inhaled COPD medication (as measured with a score of 2 or greater on a protocol-specific participant self-assessment scale of forgetting to take the medication in the last 7 days)
* Access to (and comfort with) a digital device (Desktop; Laptop; Tablet), with updated Firefox or Chrome browsers installed (or willing to download up-to-date version for the study), and daily home access to internet
* Need to have personal e-mail account that is used daily

Key Exclusion Criteria:

* Patients with asthma
* Patient with a worsening COPD episode requiring medical intervention within 4 weeks of enrolment
* Patients who have completed a pulmonary rehabilitation (PR) program in the 6 months prior to enrolment or patients who are currently in a PR program (rationale: PR programs typically include a self-management component which may interfere with study objectives)
* Planned vacation period during the study period that requires overnight stays away from home
* Major surgery performed within 6 weeks prior to enrolment or planned within 2 months after enrolment, e.g. hip replacement
* Patients prescribed inhaled COPD medications other than Spiriva Respimat plus albuterol or Stiolto Respimat plus albuterol
* Previous enrolment in study 352.2133
* Previous enrolment in this study Further exclusion criteria apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-17 (Estimated); Primary Completion 2021-07-12 (Estimated); Study Completion 2021-09-06 (Estimated)

PRIMARY OUTCOMES:
Patient interaction with TARA (engagement via usage data) | up to 3 weeks
  Data sourced from individual and amalgamated usage analytics. Data points collected from TARA Patient database / usage analytics, recording the completion with time and date stamps by the users of key sections of the TARA program. An overall score for perceived ease-of-use will be generated using the System Usability Scale (SUS) participant questionnaire
Assessment of usability issues | up to 3 weeks
  Qualitative assessment of participant's feedback on any usability issues, areas of confusion or lack of clarity whilst using TARA working prototype (version 2).
  Data sourced from participant's reports, emails and exit interviews.
Assessment of motivation and perception | up to 3 weeks
  Qualitative assessment of data sourced through the prototype and via discussion in the exit interview

SECONDARY OUTCOMES:
Percent of individuals with COPD who achieve improvements in intention (Readiness for Change) measured by the Readiness for Change Questionnaire | up to 3 weeks
Percent of individuals with COPD who achieve improvements in autonomous motivation measured by the Treatment Self-Regulation Questionnaire (TSRQ) | up to 3 weeks
Percent of individuals with COPD who achieve confidence measured by the Perceived Competence Scale; PCS) | up to 3 weeks
Percent of participants who increased adherence to once daily inhaled medication, based on Test of Adherence to Inhalers (TAI) Questionnaire | up to 3 weeks
Percent of participants who report increases in adherence to once daily inhaled medication, based on study-specific medication adherence question | up to 3 weeks
  Medication adherence question: "During the last 7 days, how many times did you forget to take your daily inhaler ?"
Percent of participants who report increases in adherence to once daily inhaled medication, based on prescription re-fill confirmation | up to 3 weeks
Percent of participants who report increases in adherence to once daily inhaled medication, based on TARA daily check-in data. | up to 3 weeks
Percent of study participants who report a reduction in COPD symptoms measured via the COPD Assessment test (CAT) | up to 3 weeks

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).For more details refer to: http://trials.boehringer-ingelheim.com/